CLINICAL TRIAL: NCT03455218
Title: Nitric Oxide Administration During Pediatric Cardiopulmonary Bypass Surgery to Prevent Platelet activation-a Single Center Pilot Study
Brief Title: Nitric Oxide Administration During Pediatric Cardiopulmonary Bypass Surgery to Prevent Platelet Activation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Mallinckrodt (Industry); Clinical & Translational Science Institute of Southeast Wisconsin (Other); Versiti Blood Health (Other)
Responsible Party: Principal Investigator, Robert Niebler, MD, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1111115-1NO in CPB 001
Record Dates: First submitted 2018-02-06; First posted 2018-03-06 (Actual); Results first posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-07

CONDITIONS: Inflammation; Platelet Dysfunction
Keywords: Cardiopulmonary Bypass; Infant; Nitric Oxide; Thrombocytopenia; Blood Platelets
MeSH Terms: conditions — Inflammation; Thrombocytopenia | interventions — Nitric Oxide; Endothelium-Dependent Relaxing Factors

STUDY DESIGN:
Intervention Model Description: Randomized, Double Blinded, Placebo Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Nitric Oxide (Experimental): 20 ppm of Nitric Oxide delivered to the oxygenator via the INOmax device for the duration of the cardiopulmonary bypass time
  Interventions: Drug: Nitric Oxide; Device: INOmax
- Placebo (Placebo Comparator): INOmax device attached to the oxygenator, but no gas is delivered through the device
  Interventions: Drug: Placebo; Device: INOmax

INTERVENTIONS:
Drug: Nitric Oxide — 20 ppm of Nitric Oxide gas delivered to the oxygenator for the duration of cardiopulmonary bypass
  Other Names: INOmax
  Arms: Nitric Oxide
Drug: Placebo — INOmax device connected to oxygenator, but no gas is delivered
  Arms: Placebo
Device: INOmax — All patients will have the INOmax device connected to the oxygenator
  Other Names: inhaled nitric oxide delivery device

SUMMARY:
Open heart surgery requires the use of a cardiopulmonary bypass (CPB) circuit. As blood flows across the artificial surfaces of the CPB circuit, platelets are activated and consumed. This activation results in a profound inflammatory reaction and need for transfusion. This reaction is intensified in younger, smaller patients undergoing longer, more complex open heart surgery. Nitric oxide is naturally released by vascular endothelial surfaces and acts as a signaling molecule which prevents platelet activation. The investigators hypothesize that the addition of the nitric oxide to the sweep gas of the oxygenator during cardiopulmonary bypass surgery will replace this natural endothelial function and thus prevent platelet activation and consumption. The investigators plan to test this hypothesis with a pilot double blinded, randomized trial of 40 patients less than a year of age undergoing cardiac surgery requiring CPB.

DETAILED DESCRIPTION:
Open heart surgery requires the use of a CPB circuit. As blood flows across the artificial surfaces of the CPB circuit, platelets are consumed (1). The investigators recently completed a prospective observational trial of neonates undergoing cardiac surgery requiring CPB. In this trial the investigators demonstrated a dramatic decrease in platelet count from baseline to intraoperatively. The platelet count rebounded with transfusion and normalized by the time of admission to the cardiac intensive care unit (CICU). Despite prophylactic transfusion of blood products to all patients, 41% experienced excessive postoperative bleeding (defined in terms of chest tube output and need for reoperation).

Further investigation by Dr. Debra Newman in her lab at the Blood Research Institute delineated the platelet defect associated with CPB in the neonates more clearly. Dr. Newman found a significant decrease in the platelet responsiveness to thrombin receptor activating protein (TRAP), thromboxane A2 analog (U46619), and collagen-related peptide (CRP). Further analysis revealed that the effect of CPB on platelet responsiveness to TRAP and U46619 is likely dependent on its effect on platelet count, whereas CPB affects platelet responsiveness to CRP independently of platelet count.

In children, postoperative blood loss and transfusion of blood products has been shown to contribute significantly to the morbidity and mortality of surgeries that require CPB (2, 3). In addition to the need for blood product replacement, the activation of platelets contributes to the intense inflammatory reaction seen in surgeries requiring CPB (4). Patients with a less intense inflammatory response post-operatively generally do better with less morbidity (5).

The oxygenator membrane surface of the CPB pump is a large contributor to the surface area of CPB circuit. As a major contributor to the surface area of the circuit and the location of the gas interface, the oxygenator is a significant contributor to the hemostatic and inflammatory stimulus of CPB. Advances in oxygenator technology have modified the surface to prevent interaction with the blood, but no artificial surface has been found to be as inert as the natural endothelium of the vasculature (5).

A major mechanism by which endothelial surfaces inhibit activation of platelets is by producing nitric oxide (6). Nitric oxide is lipophilic and traverses cellular membranes where it acts on intracellular signaling pathways in platelets to prevent platelet activation and aggregation (7). The artificial surface of the CPB pump does not produce nitric oxide and hence is devoid of this potent inhibitor of platelet activation.

In multiple experimental ex-vivo models of CPB, the addition of nitric oxide to the sweep gas of the oxygenator resulted in preserved platelet counts, preserved platelet function, and decreased markers of platelet activation (8-11).

Multiple clinical trials of nitric oxide administration during CPB have shown positive results. Chung et al. showed in a group of 41 adults undergoing coronary artery surgery requiring CPB that the addition of nitric oxide to the oxygenator resulted in a preservation of platelet numbers, a decrease in markers of platelet activation, and less post-operative blood loss (12). Checchia et al. investigated the effect of nitric oxide in a group of sixteen infants undergoing repair of tetralogy of Fallot and found the patients treated with nitric oxide had an improvement in clinical outcomes of length of stay in the intensive care unit and number of hours requiring mechanical ventilation (13). James et al. showed a 50% decrease in the incidence of low cardiac output syndrome in a randomized trial of 198 children. The effect was most profound in the younger children and those undergoing the most complex repairs (14). These patients are also the ones demonstrated to have the most intense inflammatory reaction postoperatively (15).

Despite these promising studies, several questions remain. The mechanism of platelet preservation has not been delineated. The collaboration between clinicians at Children's Hospital of Wisconsin and Dr. Newman at the Blood Center of Wisconsin has been established and has experience in investigating the effects of CPB on platelets in infants. This collaboration is poised to help define the mechanism of nitric oxide in preserving platelet function during CPB in infants. All studies to date have been single center and underpowered to investigate clinical outcomes of interest such as mortality and length of hospital stay. Dr. Niebler has begun to assemble a multi-center study team. Local data is necessary to help guide the power calculation in determining the sample size for this larger study and to demonstrate the capabilities of the local institution in leading a trial of this magnitude.

ELIGIBILITY:
Inclusion Criteria:

* Infants less than one year of age
* Undergoing cardiac surgery with the use of cardiopulmonary bypass

Exclusion Criteria:

* Prior surgery requiring CPB within the same hospitalization
* Pre-operative need for extracorporeal membrane oxygenation or mechanical circulatory support
* Known hypersensitivity to nitric oxide
* Known hemostatic or thrombotic disorder that results in an altered transfusion/anticoagulation protocol

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2019-04-20 (Actual); Study Completion 2019-05-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided
we are willing to share the IPD if requested by another investigator. Please contact the principle investigator if interested

REFERENCES:
- [Background] Despotis GJ, Avidan MS, Hogue CW Jr. Mechanisms and attenuation of hemostatic activation during extracorporeal circulation. Ann Thorac Surg. 2001 Nov;72(5):S1821-31. doi: 10.1016/s0003-4975(01)03211-8. PMID 11722116
- [Background] Chambers LA, Cohen DM, Davis JT. Transfusion patterns in pediatric open heart surgery. Transfusion. 1996 Feb;36(2):150-4. doi: 10.1046/j.1537-2995.1996.36296181928.x. PMID 8614966
- [Background] Petaja J, Lundstrom U, Leijala M, Peltola K, Siimes MA. Bleeding and use of blood products after heart operations in infants. J Thorac Cardiovasc Surg. 1995 Mar;109(3):524-9. doi: 10.1016/S0022-5223(95)70284-9. PMID 7877314
- [Background] Rinder CS, Bonan JL, Rinder HM, Mathew J, Hines R, Smith BR. Cardiopulmonary bypass induces leukocyte-platelet adhesion. Blood. 1992 Mar 1;79(5):1201-5. PMID 1371416
- [Background] Wan S, LeClerc JL, Vincent JL. Inflammatory response to cardiopulmonary bypass: mechanisms involved and possible therapeutic strategies. Chest. 1997 Sep;112(3):676-92. doi: 10.1378/chest.112.3.676. PMID 9315800
- [Background] Radomski MW, Vallance P, Whitley G, Foxwell N, Moncada S. Platelet adhesion to human vascular endothelium is modulated by constitutive and cytokine induced nitric oxide. Cardiovasc Res. 1993 Jul;27(7):1380-2. doi: 10.1093/cvr/27.7.1380. PMID 7504587
- [Background] Naseem KM, Roberts W. Nitric oxide at a glance. Platelets. 2011;22(2):148-52. doi: 10.3109/09537104.2010.522629. Epub 2010 Nov 4. PMID 21050056
- [Background] Annich GM, Meinhardt JP, Mowery KA, Ashton BA, Merz SI, Hirschl RB, Meyerhoff ME, Bartlett RH. Reduced platelet activation and thrombosis in extracorporeal circuits coated with nitric oxide release polymers. Crit Care Med. 2000 Apr;28(4):915-20. doi: 10.1097/00003246-200004000-00001. PMID 10809259
- [Background] de Graaf JC, Banga JD, Moncada S, Palmer RM, de Groot PG, Sixma JJ. Nitric oxide functions as an inhibitor of platelet adhesion under flow conditions. Circulation. 1992 Jun;85(6):2284-90. doi: 10.1161/01.cir.85.6.2284. PMID 1591842
- [Background] Konishi R, Shimizu R, Firestone L, Walters FR, Wagner WR, Federspiel WJ, Konishi H, Hattler BG. Nitric oxide prevents human platelet adhesion to fiber membranes in whole blood. ASAIO J. 1996 Sep-Oct;42(5):M850-3. doi: 10.1097/00002480-199609000-00111. PMID 8945004
- [Background] Mellgren K, Friberg LG, Mellgren G, Hedner T, Wennmalm A, Wadenvik H. Nitric oxide in the oxygenator sweep gas reduces platelet activation during experimental perfusion. Ann Thorac Surg. 1996 Apr;61(4):1194-8. doi: 10.1016/0003-4975(96)00017-3. PMID 8607682
- [Background] Chung A, Wildhirt SM, Wang S, Koshal A, Radomski MW. Combined administration of nitric oxide gas and iloprost during cardiopulmonary bypass reduces platelet dysfunction: a pilot clinical study. J Thorac Cardiovasc Surg. 2005 Apr;129(4):782-90. doi: 10.1016/j.jtcvs.2004.06.049. PMID 15821644
- [Background] Checchia PA, Bronicki RA, Muenzer JT, Dixon D, Raithel S, Gandhi SK, Huddleston CB. Nitric oxide delivery during cardiopulmonary bypass reduces postoperative morbidity in children--a randomized trial. J Thorac Cardiovasc Surg. 2013 Sep;146(3):530-6. doi: 10.1016/j.jtcvs.2012.09.100. Epub 2012 Dec 8. PMID 23228403
- [Background] James C, Millar J, Horton S, Brizard C, Molesworth C, Butt W. Nitric oxide administration during paediatric cardiopulmonary bypass: a randomised controlled trial. Intensive Care Med. 2016 Nov;42(11):1744-1752. doi: 10.1007/s00134-016-4420-6. Epub 2016 Sep 30. PMID 27686343
- [Background] Eisses MJ, Chandler WL. Cardiopulmonary bypass parameters and hemostatic response to cardiopulmonary bypass in infants versus children. J Cardiothorac Vasc Anesth. 2008 Feb;22(1):53-9. doi: 10.1053/j.jvca.2007.06.006. Epub 2007 Aug 22. PMID 18249331
- [Background] Miller BE, Mochizuki T, Levy JH, Bailey JM, Tosone SR, Tam VK, Kanter KR. Predicting and treating coagulopathies after cardiopulmonary bypass in children. Anesth Analg. 1997 Dec;85(6):1196-202. doi: 10.1097/00000539-199712000-00003. PMID 9390579
- [Background] Williams GD, Bratton SL, Riley EC, Ramamoorthy C. Coagulation tests during cardiopulmonary bypass correlate with blood loss in children undergoing cardiac surgery. J Cardiothorac Vasc Anesth. 1999 Aug;13(4):398-404. doi: 10.1016/s1053-0770(99)90210-0. PMID 10468251
- [Background] Berger JT, Holubkov R, Reeder R, Wessel DL, Meert K, Berg RA, Bell MJ, Tamburro R, Dean JM, Pollack MM; Eunice Kennedy Shriver National Institute of Child Health and Human Development Collaborative Pediatric Critical Care Research Network. Morbidity and mortality prediction in pediatric heart surgery: Physiological profiles and surgical complexity. J Thorac Cardiovasc Surg. 2017 Aug;154(2):620-628.e6. doi: 10.1016/j.jtcvs.2017.01.050. Epub 2017 Feb 10. PMID 28274558

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nitric Oxide | Placebo
Started | 18 | 22
Completed | 18 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nitric Oxide | Placebo | Total
Number analyzed (Participants) | 18 | 22 | 40
Age, Continuous [Mean (Standard Deviation); unit: Days] | 100.6 (77.7) | 112.4 (92.5) | 107.1 (85.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 9 | 13 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 13 | 19 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
Weight [Mean (Standard Deviation); unit: Kilogram] | 4.62 (1.50) | 4.80 (1.48) | 4.72 (1.47)
Known Genetic Disorder [Count of Participants; unit: Participants] | 12 | 15 | 27
STAT Category [Count of Participants; unit: Participants] — Society of Thoracic Surgery-European Association for Cardiothoracic Surgery Categorization of Surgical Complexity-graded 1, 2, 3, 4, and 5 with 1 being the most complex surgeries and 5 being the least complex surgeries. These categories are validated via the STS database to correlate with risk of mortality. To simplify reporting and randomization we designated high risk surgeries to be STAT category 1 & 2 and low risk surgeries to be STAT category 3-5.
  Participants
    STAT Category 1 & 2 | 10 | 10 | 20
    STAT Category 3-5 | 8 | 12 | 20
Total Cardiopulmonary Bypass Time [Median (Inter-Quartile Range); unit: Minutes] | 123.5 [98.8 to 155.3] | 115.0 [96 to 160.3] | 115.0 [96.5 to 158.8]
Total Aortic Cross Clamp Time [Mean (Standard Deviation); unit: Minutes] | 77.4 (40.6) | 74.1 (45.4) | 75.6 (42.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Platelet Count
Description: Change in platelet count from baseline to conclusion of cardiopulmonary bypass = (Platelet count at end of CPB) - (Platelet count prior to start of CPB)
Time Frame: From baseline to end of cardiopulmonary bypass (2-6 hours)
Measure: Mean (Standard Deviation); unit: Count of platelets
Arm/Group | Nitric Oxide | Placebo
Number analyzed (Participants) | 18 | 22
Count of platelets | -221 (107) | -242 (114)
Statistical Analysis 1: Comparison: Nitric Oxide vs Placebo; Test type: Superiority; p = 0.55, t-test, 2 sided

2. Primary Outcome: 30 Day Mortality
Description: 30 day all cause mortality
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Nitric Oxide | Placebo
Number analyzed (Participants) | 18 | 22
Participants | 0 | 0

3. Primary Outcome: Hospital Length of Stay
Description: Length of stay in the hospital following the operation
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Nitric Oxide | Placebo
Number analyzed (Participants) | 18 | 22
Days | 8 [5 to 39.3] | 16.5 [8.3 to 28.8]
Statistical Analysis 1: Comparison: Nitric Oxide vs Placebo; Test type: Superiority; p = 0.30, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Methemoglobin Level Pre-CPB
Description: Methemoglobin levels in the blood measured at baseline
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: % methemoglobin
Arm/Group | Nitric Oxide | Placebo
Number analyzed (Participants) | 18 | 22
% methemoglobin | 0.77 (0.42) | 0.99 (0.40)
Statistical Analysis 1: Comparison: Nitric Oxide vs Placebo; Test type: Superiority; p = 0.11, t-test, 2 sided

5. Primary Outcome: Methemoglobin Level-End of CPB
Description: Methemoglobin Level obtained at the end of cardiopulmonary bypass
Time Frame: 4 hours
Measure: Mean (Standard Deviation); unit: % methemoglobin
Arm/Group | Nitric Oxide | Placebo
Number analyzed (Participants) | 18 | 22
% methemoglobin | 1.56 (0.43) | 1.10 (0.43)
Statistical Analysis 1: Comparison: Nitric Oxide vs Placebo; Test type: Superiority; p = 0.002, t-test, 2 sided

6. Primary Outcome: Methemoglobin Level-ICU Admit
Description: Methemoglobin level obtained at the time of ICU Admit
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: % methemoglobin
Arm/Group | Nitric Oxide | Placebo
Number analyzed (Participants) | 18 | 22
% methemoglobin | 1.3 (0.49) | 1.08 (0.29)
Statistical Analysis 1: Comparison: Nitric Oxide vs Placebo; Test type: Superiority; p = 0.05, t-test, 2 sided

7. Secondary Outcome: Change in Platelet Response to TRAP as Measured by P-selectin Expression
Description: The P-selectin expression measured as a mean florescence was measured in platelets stimulated with thrombin receptor activating protein (TRAP) was measured at baseline and at conclusion of cardiopulmonary bypass. Mean of each assessment measured multiple times at each time point. Median change values were reported. The change in these values is the outcome measure = (Platelet response to TRAP at end of CPB) - (Platelet response to TRAP prior to CPB)
Time Frame: From baseline to end of cardiopulmonary bypass (2-6 hours)
Measure: Median (Inter-Quartile Range); unit: Florescence arbitrary units
Arm/Group | Nitric Oxide | Placebo
Number analyzed (Participants) | 18 | 22
Florescence arbitrary units | 24 [-6 to 39] | 30 [7 to 58]
Statistical Analysis 1: Comparison: Nitric Oxide vs Placebo; Test type: Superiority; p = 0.27, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Change in Platelet Response to U46619 as Measured by P-selectin Expression
Description: The P-selectin expression measured as a mean florescence was measured in platelets stimulated with U46619 was measured at baseline and at conclusion of cardiopulmonary bypass. Mean of each assessment measured multiple times at each time point. Median change values were reported. The change in these values is the outcome measure = (Platelet response to U46619 at end of CPB) - (Platelet response to U46619 prior to CPB)
Time Frame: From baseline to end of cardiopulmonary bypass (2-6 hours)
Measure: Median (Inter-Quartile Range); unit: Florescence arbitrary units
Arm/Group | Nitric Oxide | Placebo
Number analyzed (Participants) | 18 | 22
Florescence arbitrary units | 51 [38 to 64] | 40 [19 to 70]
Statistical Analysis 1: Comparison: Nitric Oxide vs Placebo; Test type: Superiority; p = 0.57, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Change in Platelet Response to CRP as Measured by P-selectin Expression
Description: The P-selectin expression measured as a mean florescence was measured in platelets stimulated with CRP was measured at baseline and at conclusion of cardiopulmonary bypass. Mean of each assessment measured multiple times at each time point. Median change values were reported. The change in these values is the outcome measure = (Platelet response to CRP at end of CPB) - (Platelet response to CRP prior to CPB)
Time Frame: From baseline to end of cardiopulmonary bypass (2-6 hours)
Measure: Median (Inter-Quartile Range); unit: Florescence arbitrary units
Arm/Group | Nitric Oxide | Placebo
Number analyzed (Participants) | 18 | 22
Florescence arbitrary units | 23 [-3 to 42] | 23 [-6 to 50]

10. Secondary Outcome: Volume of Platelet Transfusion
Description: Volume per kg of platelet transfusion given to patient from the conclusion of cardiopulmonary bypass to 48 hours post-operatively
Time Frame: 48 hours post-operatively
Measure: Median (Inter-Quartile Range); unit: mL/kg
Arm/Group | Nitric Oxide | Placebo
Number analyzed (Participants) | 18 | 22
mL/kg | 4 [0 to 25] | 9.8 [0 to 32.6]
Statistical Analysis 1: Comparison: Nitric Oxide vs Placebo; Test type: Superiority; p = 0.48, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Volume of Packed Red Blood Cell Transfusion
Description: Volume per kg of packed red blood cell transfusion given to patient from the conclusion of cardiopulmonary bypass to 48 hours post-operatively
Time Frame: 48 hours post-operatively
Measure: Median (Inter-Quartile Range); unit: mL/kg
Arm/Group | Nitric Oxide | Placebo
Number analyzed (Participants) | 18 | 22
mL/kg | 3.1 [0 to 19.1] | 0 [0 to 26.1]
Statistical Analysis 1: Comparison: Nitric Oxide vs Placebo; Test type: Superiority; p = 0.96, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Transfusion Exposures
Description: Total number of transfusion exposures for a patient from the conclusion of cardiopulmonary bypass to 48 hours post-operatively
Time Frame: 48 hours post-operatively
Measure: Median (Inter-Quartile Range); unit: Transfusions
Arm/Group | Nitric Oxide | Placebo
Number analyzed (Participants) | 18 | 22
Transfusions | 2 [1 to 4] | 3 [1 to 4]
Statistical Analysis 1: Comparison: Nitric Oxide vs Placebo; Test type: Superiority; p = 0.71, t-test, 2 sided

13. Secondary Outcome: Length of Mechanical Ventilation
Description: Time (days) spent on ventilator following the operation
Time Frame: 30 days post-operatively
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Nitric Oxide | Placebo
Number analyzed (Participants) | 18 | 22
Hours | 35.7 [0 to 111.5] | 28.2 [0 to 115.4]
Statistical Analysis 1: Comparison: Nitric Oxide vs Placebo; Test type: Superiority; p = 0.97, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Vasoactive Infusion Score
Description: Highest vasoactive infusion score (VIS) within 24 hours post-operatively. Vasoactive infusion score is based on the dose of the vasoactive infusions the patient is given VIS = Dopamine dose (μg/kg/min) + Dobutamine dose (μg/kg/min) +100 × epinephrine dose (μg/kg/min) + 10 X Milrinone dose (μg/kg/min) +10,000 × Vasopressin dose (U/kg/min) + 100 × Norepinephrine dose (μg/kg/min).
  The minimum value is 0 if the patient is not on any vasoactive medications. There is no "maximum" score as there is no "maximum" dose of vasoactive medications. Higher scores indicate that the patient is on more vasoactive medications which is generally considered worse.
Time Frame: 24 hours post-operatively
Measure: Median (Inter-Quartile Range); unit: VIS Score
Arm/Group | Nitric Oxide | Placebo
Number analyzed (Participants) | 18 | 22
VIS Score | 9 [6.3 to 16.1] | 9.5 [5.5 to 15]
Statistical Analysis 1: Comparison: Nitric Oxide vs Placebo; Test type: Superiority; p = 0.53, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Number of Subjects Requiring Extracorporeal Membrane Oxygenation
Description: Dichotomous outcome-required extracorporeal membrane oxygenation within 48 hours post-operatively
Time Frame: 48 hours post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Nitric Oxide | Placebo
Number analyzed (Participants) | 18 | 22
Participants | 1 | 1
Statistical Analysis 1: Comparison: Nitric Oxide vs Placebo; Test type: Superiority; p = 1.0, Chi-squared

16. Secondary Outcome: Hospital Cost
Description: Total hospital cost at the time of discharge
Time Frame: 6 months post-operatively
Measure: Median (Inter-Quartile Range); unit: 1000's of dollars
Arm/Group | Nitric Oxide | Placebo
Number analyzed (Participants) | 18 | 22
1000's of dollars | 137.7 [99.5 to 490.7] | 224.3 [145.0 to 283.4]
Statistical Analysis 1: Comparison: Nitric Oxide vs Placebo; Test type: Superiority; p = 0.46, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: From the start of the operation till the time of hospital discharge. All patients were observed for adverse events from the start of the operation in which they were enrolled in the study till the time of hospital discharge following the operation. This ranged from 3 to 200 days.
Description: We used the definitions of major and minor adverse events as described by the Pediatric Cardiac Critical Care Consortium Database as this is a validated method to describe adverse events in pediatric patients following cardiac surgery.
Arm/Group | Nitric Oxide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/22
Serious Adverse Events (participants affected / at risk) | 3/18 | 1/22
Other Adverse Events (participants affected / at risk) | 8/18 | 10/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitric Oxide (N=18) | Placebo (N=22)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 1 (1) — Cardiac arrest requiring cardiopulmonary resuscitation
Heart block requiring pacemaker (Cardiac disorders) | 1 (1) | 0 (0) — Heart block post-surgical requiring insertion of permanent pacemaker
Unplanned reoperation (Cardiac disorders) | 1 (4) | 0 (0) — Unanticipated return to the operating room to revise anatomical surgical repair based on residual cardiac lesion
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitric Oxide (N=18) | Placebo (N=22)
Arrhythmia requiring temporary pacemaker (Cardiac disorders) | 7 (8) | 8 (8) — Arrhythmia in the postoperative period requiring use of a temporary pacemaker. Did not require insertion of a permanent pacemaker device.
Sepsis (Infections and infestations) | 3 (3) | 1 (1) — Positive blood culture, urine culture or suspicion of systemic infection resulting in antibiotic treatment for more than 72 hours
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) — Chylous pleural effusion requiring drainage
Pulmonary hypertension (Cardiac disorders) | 2 (2) | 0 (0) — Elevation in pulmonary vascular resistance requiring medical treatment.
Seizure (Nervous system disorders) | 1 (1) | 1 (1) — Seizure requiring medical treatment or identified by electroencephalogram

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/18/NCT03455218/Prot_SAP_000.pdf